CLINICAL TRIAL: NCT04425720
Title: Use of Remote Patient Monitoring (RPM) Platform for COVID-19 Patient
Brief Title: Use of Remote Monitoring for COVID-19 Patient
Acronym: RPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-11824
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: COVID
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Of Care (Active Comparator): Patients without wearable monitoring technology undergoing routine standard of care at the hospital.
  Interventions: Other: Standard of Care
- Monitored (Experimental): Patients who are diagnosed with COVID-19 and are undergoing self-quarantine will be closely monitored using a wearable device, and shared-clinical decisions will be made based on the monitored data and patient diary
  Interventions: Device: LifeSignals Biosensor 1AX*

INTERVENTIONS:
Device: LifeSignals Biosensor 1AX* — Shared-clinical decisions will be made based on the monitored data and patient diary. Two devices will be used to monitor data, LifeSignals Biosensor 1AX* and a pulse oximeter.
  Arms: Monitored
Other: Standard of Care — This group will be treated based on standard of care at our institution.
  Arms: Standard Of Care

SUMMARY:
The central hypothesis motivating this study is that remote patient monitoring (RPM) of infectious disease patients can efficiently facilitate self-isolation. Additionally, RPM can assist in more rapid identification of patients at risk, facilitate detection of patient deterioration, and enable early interventions, all of which play a vital role in resource utilization and outcomes.

DETAILED DESCRIPTION:
Aim-I To develop and test a clinical care pathway that can be utilized in similar epidemic conditions in the future. To study this aim, the investigators will be using the COVID-19 medical surge as a condition to evaluate the framework of delivering care through remote patient monitoring. The success of this care delivery model will be evaluated on ease of model implementation, patient satisfaction, clinical outcomes, and the utilization of shared decision making.

Aim-II To evaluate remote patient monitoring for appropriate resource utilization in epidemic and pandemic conditions. To evaluate this aim, the investigators plan to compare the emergency department (ED) visits and in-patient admission of patients with and without wearable remote patient monitoring devices. Additionally, the investigators will compare the number of patients that required critical interventions (mechanical ventilation and ECMO) during the hospital stay.

Aim III To evaluate the utilization of wearable technology for upfront predictions of patients that would require in-patient admissions. To evaluate this aim, patients who are diagnosed with COVID-19 and are undergoing self-quarantine will be closely monitored using a wearable device, and shared-clinical decisions will be made based on the monitored data and patient diary. The comparison group will be patients undergoing routine standard of care at the hospital. ED visits, in-patient hospital admissions, and patient satisfaction will be the outcome measures compared between the two groups.

Aim IV To evaluate the association between early identification of critical, abnormal vital signs and the prevention of serious adverse events. To evaluate this aim, patients in the monitored group and non-monitored group will be compared for ED visits, in-patient admissions, length of hospital stay, and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 positive patient
* Does not require in-patient admission

Exclusion Criteria:

* Allergic to sensor patch
* Has implanted pacemaker
* Has excessive sweating

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leff, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, Iosifidis C, Agha R. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). Int J Surg. 2020 Apr;76:71-76. doi: 10.1016/j.ijsu.2020.02.034. Epub 2020 Feb 26. PMID 32112977
- [Background] Wilder-Smith A, Chiew CJ, Lee VJ. Can we contain the COVID-19 outbreak with the same measures as for SARS? Lancet Infect Dis. 2020 May;20(5):e102-e107. doi: 10.1016/S1473-3099(20)30129-8. Epub 2020 Mar 5. PMID 32145768
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Liu K, Fang YY, Deng Y, Liu W, Wang MF, Ma JP, Xiao W, Wang YN, Zhong MH, Li CH, Li GC, Liu HG. Clinical characteristics of novel coronavirus cases in tertiary hospitals in Hubei Province. Chin Med J (Engl). 2020 May 5;133(9):1025-1031. doi: 10.1097/CM9.0000000000000744. PMID 32044814
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Grech V. Unknown unknowns - COVID-19 and potential global mortality. Early Hum Dev. 2020 May;144:105026. doi: 10.1016/j.earlhumdev.2020.105026. Epub 2020 Mar 31. PMID 32247898 (Retraction: PMID 34120096 Early Hum Dev. 2021 Aug;159:105377)
- [Background] Goh KJ, Choong MC, Cheong EH, Kalimuddin S, Duu Wen S, Phua GC, Chan KS, Haja Mohideen S. Rapid Progression to Acute Respiratory Distress Syndrome: Review of Current Understanding of Critical Illness from Coronavirus Disease 2019 (COVID-19) Infection. Ann Acad Med Singap. 2020 Mar 16;49(3):108-118. PMID 32200400
- [Background] Liu V, Kipnis P, Rizk NW, Escobar GJ. Adverse outcomes associated with delayed intensive care unit transfers in an integrated healthcare system. J Hosp Med. 2012 Mar;7(3):224-30. doi: 10.1002/jhm.964. Epub 2011 Oct 28. PMID 22038879
- [Background] Mardini L, Lipes J, Jayaraman D. Adverse outcomes associated with delayed intensive care consultation in medical and surgical inpatients. J Crit Care. 2012 Dec;27(6):688-93. doi: 10.1016/j.jcrc.2012.04.011. Epub 2012 Jun 12. PMID 22699035
- [Background] Mokart D, Lambert J, Schnell D, Fouche L, Rabbat A, Kouatchet A, Lemiale V, Vincent F, Lengline E, Bruneel F, Pene F, Chevret S, Azoulay E. Delayed intensive care unit admission is associated with increased mortality in patients with cancer with acute respiratory failure. Leuk Lymphoma. 2013 Aug;54(8):1724-9. doi: 10.3109/10428194.2012.753446. Epub 2012 Dec 26. PMID 23185988
- [Background] Cheng PK, Wong DA, Tong LK, Ip SM, Lo AC, Lau CS, Yeung EY, Lim WW. Viral shedding patterns of coronavirus in patients with probable severe acute respiratory syndrome. Lancet. 2004 May 22;363(9422):1699-700. doi: 10.1016/S0140-6736(04)16255-7. PMID 15158632
- [Background] Weiss P, Murdoch DR. Clinical course and mortality risk of severe COVID-19. Lancet. 2020 Mar 28;395(10229):1014-1015. doi: 10.1016/S0140-6736(20)30633-4. Epub 2020 Mar 17. No abstract available. PMID 32197108
- [Background] Tian S, Hu W, Niu L, Liu H, Xu H, Xiao SY. Pulmonary Pathology of Early-Phase 2019 Novel Coronavirus (COVID-19) Pneumonia in Two Patients With Lung Cancer. J Thorac Oncol. 2020 May;15(5):700-704. doi: 10.1016/j.jtho.2020.02.010. Epub 2020 Feb 28. PMID 32114094
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Bonow RO, Fonarow GC, O'Gara PT, Yancy CW. Association of Coronavirus Disease 2019 (COVID-19) With Myocardial Injury and Mortality. JAMA Cardiol. 2020 Jul 1;5(7):751-753. doi: 10.1001/jamacardio.2020.1105. No abstract available. PMID 32219362
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Hu SB, Wong DJ, Correa A, Li N, Deng JC. Prediction of Clinical Deterioration in Hospitalized Adult Patients with Hematologic Malignancies Using a Neural Network Model. PLoS One. 2016 Aug 17;11(8):e0161401. doi: 10.1371/journal.pone.0161401. eCollection 2016. PMID 27532679
- [Background] Yancy CW. COVID-19 and African Americans. JAMA. 2020 May 19;323(19):1891-1892. doi: 10.1001/jama.2020.6548. No abstract available. PMID 32293639
- [Background] Izmailova ES, Wagner JA, Perakslis ED. Wearable Devices in Clinical Trials: Hype and Hypothesis. Clin Pharmacol Ther. 2018 Jul;104(1):42-52. doi: 10.1002/cpt.966. Epub 2018 Apr 2. PMID 29205294
- [Background] Menta AK, Subbiah IM, Subbiah V. Bringing wearable devices into oncology practice: fitting smart technology in the clinic. Discov Med. 2018 Dec;26(145):261-270. PMID 30695675
- [Background] Ip JE. Wearable Devices for Cardiac Rhythm Diagnosis and Management. JAMA. 2019 Jan 29;321(4):337-338. doi: 10.1001/jama.2018.20437. No abstract available. PMID 30633301
- [Background] Shan R, Sarkar S, Martin SS. Digital health technology and mobile devices for the management of diabetes mellitus: state of the art. Diabetologia. 2019 Jun;62(6):877-887. doi: 10.1007/s00125-019-4864-7. Epub 2019 Apr 8. PMID 30963188
- [Background] Radin JM, Wineinger NE, Topol EJ, Steinhubl SR. Harnessing wearable device data to improve state-level real-time surveillance of influenza-like illness in the USA: a population-based study. Lancet Digit Health. 2020 Feb;2(2):e85-e93. doi: 10.1016/S2589-7500(19)30222-5. Epub 2020 Jan 16. PMID 33334565

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Of Care | Monitored
Started | 150 | 150
Completed | 150 | 130
Not Completed | 0 | 20
Not completed — Withdrawal by Subject | 0 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Of Care | Monitored | Total
Number analyzed (Participants) | 150 | 130 | 280
Age, Customized [Mean (Inter-Quartile Range); unit: years]
  Average Age in Years | 65.50 [44 to 73] | 64 [58 to 74] | 65 [53 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 88 | 170
  Male | 68 | 42 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 90 | 89 | 179
  Not Hispanic or Latino | 60 | 41 | 101
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 150 | 130 | 280

OUTCOME MEASURES:

1. Primary Outcome: Number of Monitored Versus Non-Monitored In-patient Admission
Description: compare the number of in-patient admissions between the monitored and non-monitored patients
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | Monitored
Number analyzed (Participants) | 150 | 130
Participants | 8 | 9

2. Primary Outcome: How Many Subjects Needed to Visit the Emergency Department
Description: compare the number of participants who visited Emergency Department between both arms
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | Monitored
Number analyzed (Participants) | 150 | 130
Participants | 14 | 12

3. Primary Outcome: Length of Stay
Description: Length of stay of subject if hospitalized
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Of Care | Monitored
Number analyzed (Participants) | 150 | 130
days | 7 [1 to 14] | 7 [4.5 to 9.5]

4. Primary Outcome: How Many Completed the Patient Satisfaction Survey
Description: Survey given to patients who were monitored to ask about satisfaction with the program. A research associate calls enrolled subjects to determine their opinions having participated in the program.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Monitored
Number analyzed (Participants) | 130
Participants | 84

5. Primary Outcome: How Many Subjects End up Requiring Mechanical Ventilation and ECMO
Description: How often does a subject end up getting mechanical ventilation or ECMO
Time Frame: 14 days
Population: As only those monitored were surveyed, the following results only reflect one of the arms. There is no reason to conduct a satisfaction survey on individuals who received standard of care because they would not be aware of the monitoring option.
Measure: Count of Participants; unit: Participants
Arm/Group | Monitored
Number analyzed (Participants) | 130
Participants | 0

6. Primary Outcome: Serious Adverse Events
Description: events requiring extended hospital stay
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Of Care | Monitored
Number analyzed (Participants) | 150 | 130
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 17 days after admission
Description: As this is a novel pandemic, there are limited resources available for accurate identification of patients at high risk for respiratory failure and other adverse events. Subjects who were repeatedly admitted into the hospital will count as an adverse event. Death will count as a serious adverse event.
Arm/Group | Standard Of Care | Monitored
All-Cause Mortality (participants affected / at risk) | 2/150 | 1/130
Serious Adverse Events (participants affected / at risk) | 2/150 | 1/130
Other Adverse Events (participants affected / at risk) | 8/150 | 9/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Of Care (N=150) | Monitored (N=130)
Death (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Of Care (N=150) | Monitored (N=130)
Repeated Admission (Infections and infestations) | 8 (8) | 9 (9) — Subjects who were repeatedly admitted into the hospital

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04425720/Prot_SAP_000.pdf